CLINICAL TRIAL: NCT00677872
Title: An Open-Label Study to Evaluate the Safety and Efficacy of PRX-08066 in Patients With Pulmonary Hypertension and Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Epix Pharmaceuticals, Inc. (Industry)
Responsible Party: Elkan Gamzu, PhD, EPIX Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRX-08066-202
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: COPD; Pulmonary Hypertension
Keywords: Moderate to severe COPD and coincident pulmonary hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — 5-((4-(6-chlorothieno(2,3-d)pyrimidin-4-ylamino)piperidin-1-yl)methyl)-2-fluorobenzonitrile

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PRX-08066

INTERVENTIONS:
Drug: PRX-08066

SUMMARY:
A 3-month open label study to evaluate the safety and efficacy of PRX-08066 in patients with pulmonary hypertension and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women >40 years of age
* Diagnosis of COPD with an FEV1 above 20% and less than 65% of predicted normal and an FEV1-to-FVC ratio of less than 70%
* Diagnosis of pulmonary hypertension based on echocardiography within the last 6 months or by cardiac catheterization within the last 12 months
* New York Heart Association(NYHA)Class II or III
* Screening LVEF>55%, obtained by any appropriate method within 6 months of screening
* Baseline 6MWT distance>150m and <450m
* Written informed consent from each subject prior to the initiation of any study-related procedure
* Documented negative results (within 12 months)and Hepatitis B and Hepatitis C Serology

Exclusion Criteria:

* Treatment for pulmonary hypertension with epoprostenol (prostacyclin), trepostinil (Remodulin), iloprost (Ventavis), bosentan (Tracleer), ambrisentan (Letairis), sildenafil (Viagra), tadalafil (Cialis), or vardenafil (Levitra) within the 30 days prior to study entry
* Presence or history of any of the following cardiovascular co-morbidities or conditions: Un-controlled systemic hypertension at screening; unstable cardiovascular disease including intermittent atrial fibrillation or unstable angina within the 4 weeks prior to screening; amyloidosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis; history of myocardial infarction, coronary artery bypass graft surgery, or percutaneous cardiac intervention within the 3 months prior to screening; significant valvular heart disease; cerebrovascular accident or transient ischemic attack within 3 months prior to screening
* COPD exacerbation less than 1 month prior to screening
* Exercise tolerance limited by non-cardiac causes
* Clinically significant psychiatric, addictive, neurologic disease or condition
* Chronic renal impairment or renal insufficiency
* No clinically significant laboratory abnormalities
* Subjects currently being treated for PH with prostnoids, PDE-5 inhibitors and or endothelin receptor antagonist. The use of PDE-5 inhibitors "as needed" for erectile dysfunction is acceptable as long as the subject does not take the medication within 72 hours of an efficacy assessment. Other concomitant medications are allowed provided the subject has been on a stable dose regimen for at least 4 weeks prior to enrollment and the regimen continues and remains stable during the treatment and follow-up periods.
* History of nasal airway mass, septal perforation, chronic sinusitis, lidocaine allergy or current nasal passage condition that would decrease the safety or tolerability of a naso-esophageal catheter
* The subject has the presence, or history, of malignancy that required significant medical intervention within the preceding 3 months and/or is likely to result in death within the next 2 years
* The receipt of any investigational medication within 30 days prior to screening or anytime during the course of the study
* Women cannot be pregnant or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test (6-MWT)and mean pulmonary artery pressure (MPAP) utilizing right heart catheterization.

SECONDARY OUTCOMES:
Central hemodynamic and exercise capacity parameters utilizing RHC and CPET

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Pulmonary and Critical Care Unit, Boston, Massachusetts, United States